CLINICAL TRIAL: NCT04703621
Title: Daratumumab as a Treatment for Adult Immune Thrombocytopenia (The DART Study)
Brief Title: The DART Study- Daratumumab Treatment in ITP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Haukeland University Hospital (Other); Oslo University Hospital (Other); University Hospital, Akershus (Other); Henri Mondor University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RGCH005
Record Dates: First submitted 2020-12-04; First posted 2021-01-11 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-09

CONDITIONS: ITP
MeSH Terms: interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: The first 3 patients will be included in the safety run-in phase. The next 9 patients will be included in cohort 1 to receive 8 weekly injections. If the response rate is less than 100%, the next 9 patients will be included in cohort 2 to receive 8 weekly injections followed by 2 bi-weekly injections.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention ( safety run-in, cohort 1, cohort 2) (Experimental): Safety run-in( 3 patients): daratumumab once a week x 4 doses. If no worsening of thrombocytopenia can be attributed to study treatment or any other life-threatening events, the study will proceed to the main part.
  Cohort 1 ( 9 patients): daratumumab once a week x 8 doses
  If response is <100%:
  Cohort 2 ( 9 patients): daratumumab once a week x 8 doses followed by daratumumab every 2 weeks x 2 doses
  Interventions: Drug: Daratumumab Injection

INTERVENTIONS:
Drug: Daratumumab Injection — subcutaneious daratumumab administration
  Other Names: Darzalex

SUMMARY:
A multicenter clinical, open-label total dose-escalating phase II study with safety run-in to explore the clinical activity, total dosage, and safety of daratumumab in adult ITP patients who have not responded adequately or relapsed after corticosteroids and at least one second-line therapy including rituximab and/or TPO-RA.

DETAILED DESCRIPTION:
Many patients with chronic ITP require repeated or continuous medications to maintain a safe platelet count.

B-cell depletion with rituximab in ITP induces the differentiation of short-lived auto-immune plasma cells into pathogenic long-lived plasma cells in the spleen that was not present before treatment. It has been reported that refractory ITP is related to the presence of long-lived plasma cells, which are resistant to steroids and immunosuppressants, including rituximab.

These findings lead to the hypothesis that therapy directed against plasma cells may help overcome treatment resistance. At least in a proportion of patients, treatment resistance is caused by CD20 negative long-lived plasma cells.

This study aims to investigate the efficacy, the optimal number of treatments, and safety of anti-CD38 antibody daratumumab steroid-refractory or steroid-dependent in ITP patients who fail to respond to at least one previous second-line therapy, including rituximab and/ or TPO agonist.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years.
2. Primary ITP with a platelet count of ≤30x109/L measured within 2 weeks prior to inclusion with failure to achieve response or relapse after corticosteroid therapy, and at least one second-line therapy including rituximab (last infusion ≥ 24 weeks before study inclusion) and/or TPO-RA. The dose of steroids or/and TPO-RAs (romiplostim, eltrombopag and avatrombopag) has not been changed during the last 2 weeks preceding the inclusion. For the safety run-in phase, a platelet count of 15-30x 109/L will be required.
3. Signed and dated written informed consent.
4. Females of child-bearing potential accepting to follow effective contraceptive methods for at least 24 weeks following the administration of first daratumumab injection. A man who has not had a vasectomy and who is sexually active with a woman of childbearing potential must agree to use a barrier method of birth control e.g., a condom with spermicidal foam/film/gel/cream/suppository, and all men must also not donate sperm during the study and for 3 months following discontinuation of Daratumumab

Exclusion Criteria:

1. Patients with active bleeding during the last 7 days prior to inclusion. Active bleeding is defined as any clinically overt hemorrhage (including radiologically diagnosed bleeding) with ongoing hemoglobin fall or bleeding requiring immediate intervention.
2. Pregnancy or lactation.
3. Surgery planned within the 3 next months.
4. Secondary ITP: ITP associated with lymphoma, chronic lymphocytic leukemia, drug induced or ITP secondary to autoimmune disorders such as systemic lupus erythematosus, rheumatoid arthritis, antiphospholipid syndrome, common variable immune deficiency, human immunodeficiency virus, or hepatitis C.
5. Concomitant autoimmune hemolytic anemia.
6. Known allergy and/or sensitivity or contraindication to daratumumab.
7. Current active malignancy likely to require chemotherapy or surgical treatment during the study period or within one year after the start of the study treatment.
8. Patients with history of poor compliance or history of alcohol/drug abuse or excessive alcohol beverage consumption that would interfere with the ability to comply with the study protocol, or current or past psychiatric disease that might interfere with the ability to comply with the study protocol or give informed consent.
9. Patient unable to attend all the visits planned for the trial.
10. Positive at screening for hepatitis B virus (HBV) surface and core antibodies unrelated to vaccination:

    * patients with positive HBV surface antigen (HbsAg) are not eligible
    * patients who are HbsAg negative and HBV core antigen antibody positive (HBcAb) will be tested for HBV surface antibody (HBsAb) and HBV DNA. If HBsAb titer is >1000 IU/ml, patients may be enrolled. Monthly HBV DNA monitoring will be required while on treatment and for the 6 months after the last dose of the study drug.
    * patients who are HBcAb positive, HBsAg negative with HBsAb titer <100 IU/ml or negative, are not eligible.
11. Known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is required for participants suspected of having COPD.
12. Known moderate or severe persistent astma within the past 2 years, uncontrolled asthma of any classification.
13. Patient participating in another clinical trial with an investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
to evaluate of response after daratumumab treatment | 12-16 weeks
  Response defined as platelet count ≥50 x109/L in 2 measurements (taken at least 24 hours apart) during week 12 for safety run-in cohort 1 and during week 16 for cohort 2 (after first study drug injection) without having received rescue therapy, having had dose increment of TPO-RA or corticosteroids during the study period.
safety of daratumumab | 24 weeks
  incidence, severity and relationship of treatment emergent adverse events

SECONDARY OUTCOMES:
duration of respons (DOR) | 12-16 weeks
  duration of sustained platelet count ≥50x109/L without having received any platelet elevating therapy or having had dose increment of TPO-RA and/or corticosteroids
time to treatment failure (TTF) | minimum 24 weeks
  time with platelet count≥ 50x109/L from 4 weeks after the last daratumumab injection to the first platelet count <30x109/L of two counts taken in two consecutive measurements at least 24 hours apart, or administration of any platelet elevating therapy after achieving response
measurement of HRQoL and fatigue | 24 weeks
  measurement of HRQoL and fatigue using SF36 and MFI-20 questionnaire before daratumumab therapy, at week 8 for safety run-in, at week 12 for cohort 1, at week 16 for cohort 2 and at study week 24 for all patients in the study. Assess of difference in HRQoL and fatigue between non-responders and responders prior to and after daratumumab treatment
measurements of antibodies | 24 weeks
  level of anti-GPIIb/IIIa and Ib antibodiesbefore daratumumab therapy and at study week 24 ( only Norwegian centers)
analysis of platelet bound antibodies and functional testing of immunocompetent cells | 24 weeks
  analysis of platelet bound antibodies and functional testing of immunocompetent cells in peripheral blood and bone marrow before daratumumab therapy and at study week 24 ( only Norwegian centers)
measurements of various subsets of immunocompetent cells | 24 weeks
  characterization of various subsets of immunocompetent cells in the bone marrow and blood before daratumumab therapy and at study week 24(only Norwegian centers)
correlation between response and changes in antibody levels or of immunocompetent cells. | 24 weeks
  identify whether or not changes to antibody levels or of immunocompetent cells correlate with clinical response ( only Norwegian centers)

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Ghanima, PhD, Principal Investigator — Ostfold Hospital Trust
Locations (6):
- Odense University Hospital, Odense, Denmark
- Henri Mondor University Hospital, Créteil, France
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Ostfold Hospital Trust, Grålum
  - Akershus University Hospital, Oslo
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsykunova G, Holme PA, Tran HTT, Frederiksen H, Tjonnfjord E, Munthe LA, Drivet E, Kared H, Sorvoll IH, Ahlen MT, Mahevas M, Michel M, Bussel J, Kuter DJ, Anderson Tvedt TH, Ghanima W. Safety and efficacy of daratumumab in immune thrombocytopenia. Blood Adv. 2026 Jan 13;10(1):143-154. doi: 10.1182/bloodadvances.2025017279. PMID 40763272